CLINICAL TRIAL: NCT05187650
Title: Effectiveness of a Powered Exoskeleton Combined With Functional Electric Stimulation for Patients With Chronic Spinal Cord Injury: a Randomized Controlled Trial
Brief Title: Effectiveness of a Powered Exoskeleton Combined With FES for Patients With Chronic SCI: a RCT
Acronym: Ekso-FES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Widmer (Network)
Responsible Party: Sponsor-Investigator, Mario Widmer, Principal Investigator, Swiss Paraplegic Research, Nottwil
Organization: Swiss Paraplegic Research, Nottwil (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-08
Record Dates: First submitted 2021-11-16; First posted 2022-01-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Gait Disorders, Neurologic
Keywords: SCI; Functional Electrical Stimulation; Exoskeleton; Robotic device; Robotic overground gait training
MeSH Terms: conditions — Spinal Cord Injuries; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: assessor-blinded, exploratory, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to treatment allocation and study participants will be instructed not to talk to assessors about their treatment within the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ekso and FES (Experimental): Participants will train for 8 weeks, 3 times per week (i.e. 24 sessions in total) for 30 minutes effective training time per session using the EksoNR powered exoskeleton combined with gait-synchronized FES using the FES RehaMove2.
  Interventions: Device: Ekso (EksoNR, Ekso Bionics); Device: FES (RehaMove2, Hasomed)
- Ekso without FES (Active Comparator): Participants will train for 8 weeks, 3 times per week (i.e. 24 sessions in total) for 30 minutes effective training time per session using the EksoNR powered exoskeleton without applying FES.
  Interventions: Device: Ekso (EksoNR, Ekso Bionics)

INTERVENTIONS:
Device: Ekso (EksoNR, Ekso Bionics) — The EksoNR is a powered exoskeleton designed to be used in a rehabilitation setting. The device meets the provision of the Council Directive 93/42/EEC concerning medical devices and is used for gait training in neurorehabilitation.
Device: FES (RehaMove2, Hasomed) — RehaMove 2 sends electrical impulses via electrodes to nerves to evoke muscle contraction. The device meets the provision of the Council Directive 93/42/EEC concerning medical devices.
  Arms: Ekso and FES

SUMMARY:
While there are a number of prospective studies evaluating powered exoskeletons in SCI patients, to date, not a single well-designed, randomized clinical trial has been published. However, there is evidence for beneficial effects of over-ground exoskeleton therapy on walking function post-intervention from a meta-analysis on non-randomized, uncontrolled studies. Functional electrical stimulation (FES), on the other hand, is a common and established method for the rehabilitation of persons with SCI and has been demonstrated to be beneficial in, e.g., improving muscle force, power output and endurance.

Combining FES and overground robotic therapy within the same therapy session could potentially merge and potentiate the effects of each separate treatment, making it a very powerful and efficient therapy method. Up to date, however, comparative studies evaluating benefits of this combined approach (i.e., powered exoskeleton and FES) to robotic therapy without FES are missing.

DETAILED DESCRIPTION:
Paraplegia is a serious event that leads to a complete or partial loss of motor, sensory and vegetative functions. Regaining of gait, balance and mobility are important priorities for persons with a spinal cord injury (SCI). In the last decade the technological development of exoskeletons allowed persons with SCI getting closer to their desired goal. Wearable robotic exoskeletons are motorized orthoses that facilitate untethered standing and walking over ground. Supporting multiple step repetitions while having full weight bearing on the body, these devices represent a task-specific and -oriented training approach for rehabilitation of gait function after SCI. However, in cases where rehabilitation of gait function is not the aim, the need to target secondary health problems associated with SCI like pain, spasticity, bowel and bladder function can still be a rationale for engaging in exoskeleton training.

Another well-established technique for the treatment of such secondary health problems is functional electrical stimulation (FES). FES is a common and established method for the rehabilitation of persons with spinal cord injury. Several studies have documented positive effects of FES like, e.g., avoiding disuse and denervation atrophy, improving muscle force, power output and endurance, changing muscle fibre type, increasing cross sectional area of muscles, increasing muscle mass, activation of nerve sprouting, motor learning and reducing spasticity. In addition, FES has been shown to improve bladder, bowel and sexual function, cardiovascular fitness (by increasing aerobic capacity), reduce body fat mass and prevent and treat pressure ulcers by increasing muscular blood flow. Moreover, FES treatment has also been shown to have an impact on body function by improving lower limb function as well as trunk stability and function.

The power elicited by the muscle through electrical stimulation can be used for locomotion. To do so, undesired limb motion is often restricted by passive orthoses or pedals in order to efficiently use the muscle contraction from the user to safely provide the power for forward propulsion. The usefulness of such systems, however, is often limited due to the rapid initiation of muscle fatigue. This is one reason (amongst others) why hybrid FES-robotic solutions have been developed, which supplement the power produced by electrical stimulation with motorized assistance. This approach reduces the power that needs to be produced by the muscles, allowing for FES application for longer training sessions before fatigue occurs. By doing so, such hybrid powered exoskeletons offer the physiological health benefits similar to FES cycling, while simultaneously enhancing the user's mobility. The addition of FES to a powered exoskeleton also synergistically reduces the motor torques of the device, reducing battery drain and therefore increasing the maximum range of the exoskeleton.

While it sounds perfectly reasonable, from a technical and physiological perspective, to combine powered exoskeletons and FES to such hybrid bionic systems, there is only anecdotal evidence for their clinical usefulness and efficacy in patients with SCI. Here the investigators propose a randomized controlled trial investigating the effect of the combined application of the EksoNR powered exoskeleton (Ekso Bionics, Richmond, CA, USA) and FES (FES RehaMove2, Hasomed, Magdeburg, Germany) compared to Ekso therapy alone on functional outcomes and secondary health parameters.

ELIGIBILITY:
Inclusion Criteria:

* chronic, incomplete SCI (> 1 year, AIS B-D)
* traumatic or non-traumatic lesion
* capacity to stand up and perform a 10MWT with or without medical aids
* partially wheelchair dependent
* intact lower motoneuron on the segmental innervation level of M. glutaeus maximus, Mm. ischiocrurales, M. tibialis anterior and M. quadriceps (to guarantee the stimulability with FES)

Exclusion Criteria:

* Exoskeleton device related contraindications: > 100 kg body weight; Body height: < 155 cm or > 190 cm; pelvic width: > 46 cm
* orthopedic limitations (acute fractures of the lower limb)
* contractures
* heterotrophic ossification
* spasticity (modified Ashworth Scale >3)
* skin injuries of the lower limbs in areas where the skin has contact with the exoskeleton
* Unstable circulation (unable to stand for at least 10 minutes)
* acute deep vein thrombosis
* pregnancy (tested in women of childbearing age (15 - 49 years))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
change in preferred walking speed from baseline (Visit 1) to post-training (Visit 2) as measured by using the 10MWT | within 3 days post-training
  The 10MWT is a quantitative measurement of lower extremity function. Patients are instructed to walk 10 meters at their preferred speed. Time is measured while the individual walks the set distance (10 meters). The distance covered is divided by the time it took the individual to walk that distance.

SECONDARY OUTCOMES:
change from baseline (Visit 1) in preferred walking speed, measured by the 10MWT, at Visit 3 | 3 months post intervention
  The 10MWT is a quantitative measurement of lower extremity function. Patients are instructed to walk 10 meters at their preferred speed. Time is measured while the individual walks the set distance (10 meters). The distance covered is divided by the time it took the individual to walk that distance.
Changes from baseline at Visit 2 and Visit 3 in maximal walking speed measured by the 10MWT | within 3 days post-training, 3 months post intervention
  The 10MWT is a quantitative measurement of lower extremity function. Patients are instructed to walk 10 meters at their preferred speed. Time is measured while the individual walks the set distance (10 meters). The distance covered is divided by the time it took the individual to walk that distance.
Changes from baseline at Visit 2 and Visit 3 in gait function as measured by the Walking Index for Spinal Cord Injury II (WISCI II) | within 3 days post-training, 3 months post intervention
  WISCI is an ordinal scale that is used in clinical trials as a tool to asses walking function. It captures the extent and nature of assistance a person with SCI requires to walk. This assessment index includes a rank ordering along a dimension of impairment, from the level of most severe impairment (level 0) to least severe impairment (level 20). The level is based on the use of devices, braces and physical assistance of one or more persons. The ranking of severity is based on the severity of impairment and not on functional independence in the environment.
Changes from baseline at Visit 2 and Visit 3 in endurance as measured by the 6 Minute Walk Test (6mWT) | within 3 days post-training, 3 months post intervention
  The 6mWT is a sub-maximal test that is used as a global and easy indicator of the loco-motor performance. Individuals are instructed to walk as far as possible during 6 minutes, taking rests whenever required. The distance covered and the number/time of rests required are recorded.
Changes from baseline at Visit 2 and Visit 3 in balance function as measured by the Mini-Balance Evaluation Systems Test (Mini-BESTest) | within 3 days post-training, 3 months post intervention
  The Mini-BESTest is a 14-item test which targets dynamic balance by assessing 4 subsystems influencing balance control: anticipatory postural adjustments, postural responses, sensory orientation and balance during gait. Items are scored on an ordinal scale ranging from 0 to 2 (0=unable, 2=normal), with a total score of 28 points.
Changes from baseline at Visit 2 and Visit 3 in the standing balance assessment using the zebris pressure distribution measurement platform (zebris Medical GmbH, Isny, Germany) | within 3 days post-training, 3 months post intervention
  Patients stand upright with feet positioned in the outline of the force-plate, keeping their eyes open/closed and looking forward during the entire test. The system records the path of the centre of pressure (COP) and calculates the traveled distance, the average speed and the area of the 95% confidence ellipse of the COP during the measurement.
Changes from baseline at Visit 2 and Visit 3 in strength using the Medical Research Council Manual Muscle Test (MRC MMT) | within 3 days post-training, 3 months post intervention
  The MRC MMT is a standardized set of assessments to measure muscle strength. The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle (0=no contraction, 5=normal power).
Changes from baseline at Visit 2 and Visit 3 in Quality of Life will be assessed according to the International SCI Quality of Life Basic Data Set | within 3 days post-training, 3 months post intervention
  Quality of Life will be assessed according to the International SCI Quality of Life Basic Data Set.
Training duration in the Exoskeleton | week 1 to week 8
  The training duration in the Exoskeleton in minutes will be automatically analysed and documented by the Ekso operating software (Ekso Pulse).
Training intensity in the Exoskeleton | week 1 to week 8
  Intensity of the training will be automatically analysed and documented as steps per minutes by the Ekso operating software (Ekso Pulse).
Training volume in the Exoskeleton | week 1 to week 8
  Training volume will be automatically analysed and documented as number of steps executed for the training duration.
Cardio-respiratory measurement | week 2, week 8
  Participants will undergo an analysis of the cardio-respiratory demand of the respective therapy method using the K5 wearable metabolic system (COSMED).

OTHER OUTCOMES:
Participant characteristics | 3 months post intervention
  Participant characteristics will be collected according to the International SCI Core Data Set.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Widmer, PhD, Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shackleton C, Evans R, Shamley D, West S, Albertus Y. Effectiveness of over-ground robotic locomotor training in improving walking performance, cardiovascular demands, secondary complications and user-satisfaction in individuals with spinal cord injuries: A systematic review. J Rehabil Med. 2019 Oct 29;51(10):723-733. doi: 10.2340/16501977-2601. PMID 31511902
- [Background] Spungen AM, Bauman WA, Biswas K, Jones KM, Snodgrass AJ, Goetz LL, Gorman PH, Kirshblum S, Sabharwal S, White KT, Asselin PK, Morin KG, Cirnigliaro CM, Huang GD. The design of a randomized control trial of exoskeletal-assisted walking in the home and community on quality of life in persons with chronic spinal cord injury. Contemp Clin Trials. 2020 Sep;96:106102. doi: 10.1016/j.cct.2020.106102. Epub 2020 Aug 12. PMID 32800962
- [Background] Gater DR Jr, Dolbow D, Tsui B, Gorgey AS. Functional electrical stimulation therapies after spinal cord injury. NeuroRehabilitation. 2011;28(3):231-48. doi: 10.3233/NRE-2011-0652. No abstract available. PMID 21558629
- [Background] Gorgey AS, Harnish CR, Daniels JA, Dolbow DR, Keeley A, Moore J, Gater DR. A report of anticipated benefits of functional electrical stimulation after spinal cord injury. J Spinal Cord Med. 2012 Mar;35(2):107-12. doi: 10.1179/204577212X13309481546619. PMID 22525324
- [Background] Ditunno PL, Patrick M, Stineman M, Ditunno JF. Who wants to walk? Preferences for recovery after SCI: a longitudinal and cross-sectional study. Spinal Cord. 2008 Jul;46(7):500-6. doi: 10.1038/sj.sc.3102172. Epub 2008 Jan 22. PMID 18209742
- [Background] Kozlowski AJ, Bryce TN, Dijkers MP. Time and Effort Required by Persons with Spinal Cord Injury to Learn to Use a Powered Exoskeleton for Assisted Walking. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):110-21. doi: 10.1310/sci2102-110. Epub 2015 Apr 12. PMID 26364280
- [Background] Zeilig G, Weingarden H, Zwecker M, Dudkiewicz I, Bloch A, Esquenazi A. Safety and tolerance of the ReWalk exoskeleton suit for ambulation by people with complete spinal cord injury: a pilot study. J Spinal Cord Med. 2012 Mar;35(2):96-101. doi: 10.1179/2045772312Y.0000000003. Epub 2012 Feb 7. PMID 22333043
- [Background] Ha KH, Murray SA, Goldfarb M. An Approach for the Cooperative Control of FES With a Powered Exoskeleton During Level Walking for Persons With Paraplegia. IEEE Trans Neural Syst Rehabil Eng. 2016 Apr;24(4):455-66. doi: 10.1109/TNSRE.2015.2421052. Epub 2015 Apr 23. PMID 25915961
- [Background] Charlifue S, Post MW, Biering-Sorensen F, Catz A, Dijkers M, Geyh S, Horsewell J, Noonan V, Noreau L, Tate D, Sinnott KA. International Spinal Cord Injury Quality of Life Basic Data Set. Spinal Cord. 2012 Sep;50(9):672-5. doi: 10.1038/sc.2012.27. Epub 2012 Mar 27. PMID 22450884